CLINICAL TRIAL: NCT04964362
Title: The Impact of Injustice Appraisals on Psychosocial Outcomes Following Spinal Cord Injury: A Longitudinal Study
Status: Active, not recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PMR-2021-30041
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with Spinal Cord Injury: Individuals with recent spinal cord injuries, both veterans and civilians, will be followed for 1 year for inquiry into injustice appraisals.

SUMMARY:
The primary objectives of this study are to: (1) determine the longitudinal course and impact of injury-related injustice appraisals among civilians and Veterans who have recently acquired a spinal cord injury (SCI), and (2) use qualitative inquiry to gain a rich, contextual understanding of appraisals of injustice during the first year after acquired SCI. The long-term goal of this research is to inform the development of new treatment approaches targeting appraisals of injustice.

DETAILED DESCRIPTION:
At present, there are no interventions that specifically target appraisals of injustice, and there is limited research upon which to recommend clinical interventions to mitigate the impact of injustice appraisals on rehabilitation outcomes. Treatment techniques currently being used within multidisciplinary rehabilitation programs do not yield clinically meaningful reductions in perceptions of injustice. Findings from the proposed study will inform the development of interventions targeting injustice appraisals and associated sequelae. Given the lack of research in this domain, as well as the absence of interventions to address injustice appraisals following injury, the proposed study will make a significant contribution to our current understanding of mechanisms that impact psychosocial and functional outcomes following spinal cord injury to inform future interventions.

ELIGIBILITY:
Inclusion Criteria:

* Have acquired a spinal cord injury (SCI) in the past 6 months
* Admitted for first inpatient rehabilitation hospitalization

Exclusion Criteria:

* SCI without neurological impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans and civilians who have recently acquired a spinal cord injury and are hospitalized for inpatient rehabilitation through the University of Minnesota Health System, Jefferson-affiliated rehabilitation hospitals, the Minneapolis VA Health Care System, and the Richmond VA Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Injustice Experience Questionnaire (IEQ) Score | 12 months
  Injustice appraisals will be measured via the IEQ. The IEQ asks participants to rate 12 statements describing different thoughts and feelings they may experience when they think about their injuries on a 5-point scale from 0 (never) to 4 (all the time). Scores range from 0 to 48; higher scores represent greater appraisals of injustice. The IEQ has strong psychometric properties among individuals with persistent musculoskeletal pain, among an acute trauma sample, and within rehabilitation settings. The IEQ will be collected at inpatient rehabilitation/acute phase (baseline), 6 months post-discharge/sub-acute phase (T1), and 12 months post- discharge/chronic phase (T2).
The Appraisals of Disability Primary and Secondary Scale- Short Form (ADAPSSsf) Score | 12 months
  The ADAPSSsf will be used to assess appraisals of disability. The ADAPSSsf is a 6-item self-report survey of people's thoughts about their spinal cord injuries.
  Each item on the ADAPSSsf represents a subscale: Fearful Despondency, Overwhelming Disbelief, Determined Resolve, Growth and Resilience, Negative Perceptions, and Personal Agency. Items are rated on a 6-point scale (strongly disagree to strongly agree) and summed (items 3, 5, and 6 are reverse coded), with higher scores representing less adaptive appraisals. The ADAPSS was developed and validated for use in the spinal cord injury population. The ADAPSSsf will be collected at inpatient rehabilitation/acute phase (baseline), 6 months post-discharge/sub-acute phase (T1), and 12 months post- discharge/chronic phase (T2).
Patient Health Questionnaire-8 (PHQ-8) Score | 12 months
  The PHQ-8 asks participants to rate how often they have been bothered by eight symptoms of depression over the past two weeks on a 0 (not at all) to 3 (nearly every day) scale. Scores on the PHQ-8 are summed to indicate the severity of depression symptoms, with higher scores indicating increasing severity. The PHQ-8 is a valid and reliable measure to assess depression in persons with spinal cord injury. The PHQ-8 will be collected at inpatient rehabilitation/acute phase (baseline), 6 months post-discharge/sub-acute phase (T1), and 12 months post- discharge/chronic phase (T2).
Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) Score | 12 months
  The PCL-5 is a 20- item self-report measure assessing symptoms of PTSD. Participants rate how bothered they have been by each of the 20 items in the past month on a 5-point scale ranging from 0 (not at all) to 4 (extremely). Scores range from 0-80, with higher scores indicating greater severity of PTSD symptoms. The PCL-5 is psychometrically sound in civilians and veterans. The PCL-5 will be collected at inpatient rehabilitation/acute phase (baseline), 6 months post-discharge/sub-acute phase (T1), and 12 months post- discharge/chronic phase (T2).
Spinal Cord Injury-Functional Index/Assistive Technology Short Forms (SCI-FI/AT) Score | 12 months
  The SCI-FI/AT assesses functional impairment in four domains:
  basic mobility (9 items), self-care (9 items), fine motor (9 items), and ambulation (8 items). For each item, participants select the response that best describes their ability to do each activity without help from another person but using the equipment or devices they usually use. Items are rated from 0 (unable to do so) to 4 (without any difficulty). Summed raw scores are transformed into T scores in each domain. The SCI-FI/AT has excellent psychometric properties. The SCI-FI/AT will be collected at inpatient rehabilitation/acute phase (baseline), 6 months post-discharge/sub-acute phase (T1), and 12 months post- discharge/chronic phase (T2).
International Spinal Cord Injury Pain Basic Data Set (ISCIPBDS) | 12 months
  The ISCIPBDS asks participants if they have experienced pain in the past seven days. If pain was experienced, three 11-point Likert scale questions pertaining to pain interference are asked, ranging from no interference to extreme interference. Total scores range from 0 to 30, and higher scores indicate greater interference due to pain.The ISCIPBDS is appropriate for the evaluation of pain among community-dwelling individuals with SCI. The ISCIPBDS will be collected at inpatient rehabilitation/acute phase (baseline), 6 months post-discharge/sub-acute phase (T1), and 12 months post- discharge/chronic phase (T2).
The International Spinal Cord Injury Quality of Life Basic Data Set (ISCIQOLBDS) | 12 months
  The ISCIQOLBDS assesses three aspects of QoL: satisfaction with general QoL (overall well-being), satisfaction with physical health, and satisfaction with psychological health. Each factor is rated on a 0-10 scale from 0 (completely dissatisfied) to 10 (completely satisfied). Higher scores on each factor indicate higher QoL in that domain. The ISCIQOLBDS demonstrates good psychometric populations. The ISCIQOLBDS will be collected at inpatient rehabilitation/acute phase (baseline), 6 months post-discharge/sub-acute phase (T1), and 12 months post- discharge/chronic phase (T2).
State-Trait Anger Expression Inventory-2 (STAXI-II) Score | 12 months
  The STAXI-II includes four subscales: state (7 items), trait (5 items), expression (4 items), and anger inhibition (4 items). The state subscale reflects the intensity of an individual's feelings of anger at the time of testing; the trait subscale assesses a person's general predisposition to become angry. Anger inhibition items reflect the frequency with which individuals attempt to suppress feelings of anger, whereas anger expression items gauge how often anger is outwardly expressed. The STAXI-II has been used in previous spinal cord injury research and demonstrates excellent psychometric properties across use with outpatient, inpatient, and rehabilitation populations. The STAXI-II will be collected at inpatient rehabilitation/acute phase (baseline), 6 months post-discharge/sub-acute phase (T1), and 12 months post- discharge/chronic phase (T2).
Qualitative Interview | 12 months
  Qualitative interviews will be conducted with a subset of individuals to explore injustice appraisals during inpatient rehabilitation and 12 months post-rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley Monden, PhD, Principal Investigator — University of Minnesota Medical School Department of Rehabilitation Medicine
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No